CLINICAL TRIAL: NCT04052334
Title: A Phase I Trial of Lymphodepletion Plus Adoptive Cell Therapy With High-Dose IL-2 in Adolescent and Young Adult Patients With Soft Tissue Sarcoma
Brief Title: Lymphodepletion Plus Adoptive Cell Therapy With High Dose IL-2 in Adolescent and Young Adult Patients With Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Iovance Biotherapeutics, Inc. (Industry); The V Foundation for Cancer Research (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19837; 1K08CA252642-01 (NIH)
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Sarcoma
Keywords: Soft Tissue Sarcoma; Adoptive Cell Therapy
MeSH Terms: conditions — Sarcoma | interventions — Interleukin-2; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Infusion of Tumor-infiltrating lymphocyte (Experimental): Participants will undergo tumor resection from which the tumor infiltrating lymphocyte (TIL) product will be generated. All participants will receive nonmyeloablative lymphodepleting chemotherapy with cyclophosphamide and fludarabine to enhance T-cell persistence and effectiveness in vivo. Cyclophosphamide will be administered at 60 mg/kg/day IV in 250 mL normal saline (NS). Fludarabine will then be infused at 25 mg/m^2 intravenous piggyback (IVPB). All participants will receive not less than 10^9, and up to 1x10^12 T cells in ≥250 mL NS as an inpatient by intravenously (IV).
  Eight (8) to sixteen (16) hours after completing the T cell infusion, all participants will receive high-dose interleukin-2 (IL-2) on an inpatient basis at the standard dose of 600 000 IU/kg as an intravenous bolus over an approximate 15-minute period every 8 to 16 hours for up to 15 doses on days 1 to 5, as tolerated.
  Interventions: Drug: TIL; Drug: Interleukin-2; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: TIL — Participants will receive an infusion of Tumor-infiltrating lymphocytes (TIL) after tumor resection and TIL product is generated.
  Other Names: Tumor-infiltrating lymphocytes
Drug: Interleukin-2 — Participants will receive Interleukin-2 (IL-2) 600 000 IU/kg intravenously (IV) bolus (about 15 minutes) every 8 to 16 hours for up to 15 doses, beginning approximately 8 to 16 hours after T-cell infusion.
  Other Names: IL-2
Drug: Fludarabine — Participants will receive an intravenously (IV) infusion of Fludarabine 25 mg/m2 for approximately 30 minutes for 5 days, prior to T-Cell infusion
  Other Names: Fludara
Drug: Cyclophosphamide — Participants will receive Cyclophosphamide 60 mg/kg/day intravenously (IV) in 250 mL normal saline (NS) over approximately 2 hours, 7 days prior to T-Cell infusion
  Other Names: Cytoxan; Neosar

SUMMARY:
This is a single-arm trial that will evaluate the safety and feasibility of the Tumor-infiltrating lymphocyte (TIL) treatment and the persistence of TIL survival in vivo following treatment

ELIGIBILITY:
Inclusion Criteria:

* Participants must fulfill all of the following criteria to be eligible for the study at the time of tumor resection and initiation of TIL expansion.
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Participants must have metastatic, high-grade soft tissue sarcoma, all subtypes will be eligible
* Residual measurable disease after resection of target lesion(s) for TIL growth
* Eastern Cooperative Oncology Group (ECOG) 0 to 1. ECOG performance status of 0 to 1 will be inferred if the patient's level of energy is ≥ 50% of baseline.
* Participants must have progressed on at least one prior standard of care treatment regimen for metastatic disease.
* A negative pregnancy test (urine or serum) must be documented at screening for women of childbearing potential.
* A MUGA scan (ejection fraction > 50% is required) ≤ 6 months prior to lymphodepletion.
* Pulmonary function tests should be completed ≤ 6 months prior to lymphodepletion and forced expiratory volume (FEV1) > 65% or FVC > 65% of predicted are required
* Adequate renal, hepatic, and hematologic function, including creatinine of ≤ 1.7 gm/dL, total bilirubin ≤ 2.0 mg/dL, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dL, AST and ALT of less than 3 X institutional upper limit of normal, hemoglobin of 8 gm/dL or more, white blood cells of 3000 per mm^3 and total granulocytes of 1000 per mm^3 or more, and platelets of 100 000 per mm^3 or more.
* Participants must have a positive screening EBV antibody titre on screening test.
* Participants that have had previously grown sterile, validated TILs under good manufacturing practice conditions meeting the above criteria are eligible using the previously established TIL product stored in the Cell Therapies Core facility for up to 2 years after harvesting.
* Unless surgically sterile by bilateral tubal ligation or vasectomy of partner(s), the participant agrees to continue to use a method of contraception throughout the study such as: barrier (i.e. condom, diaphragm), hormonal, IUD, or sponge plus spermicide.
* Prothrombin time (PT) and partial thromboplastin time (PTT) within 1.5 times the institutional upper limit of normal
* Participants with echocardiogram (EKG) within 14 days of initiation of chemotherapy demonstrating no new rhythm, axis, or ST segment If new ST changes are present, patients may be included if cardiac stress test indicates no evidence of inducible cardiac ischemia.
* Urinalysis within 14 days demonstrating no evidence of a urinary tract infection.
* Participants with evidence of ongoing disease regression that is attributed to a therapy that is not part of the trial and that was administered after TIL harvest and expansion but prior to adoptive transfer of TILs should continue on prior therapy and may be treated with TIL only if their disease is stable or there is evidence of progressive disease. In this event as described above, the TIL will be frozen and stored for future use, in the event of progression, prior to the rapid expansion step.

Exclusion Criteria:

* Participants with active systemic infections requiring intravenous antibiotics, coagulation disorders, or other major medical illnesses of the cardiovascular, respiratory, or immune system are excluded.
* Participants that have completed a chemotherapy regimen given with the intent of lymphodepletion or cellular immunotherapy which included non-myeloablative lymphodepletion strategy.
* Participants testing positive for HIV titer, hepatitis B surface antigen, human T-cell leukemia-lymphoma virus (HTLV) I or II antibody, or both rapid plasma regain (RPR) and fluorescent treponemal antibody (FTA) are excluded. Participants with hepatitis C antibody must have a negative (undetectable) viral load by polymerase chain reaction (PCR).
* Participants who are pregnant or nursing are excluded.
* Participants needing chronic immunosuppressive systemic steroids are excluded
* Participants with autoimmune diseases that require immunosuppressive medications are excluded
* Presence of a significant psychiatric disease, which in the opinion of the principal investigator or his designee, would prevent adequate informed consent or render immunotherapy unsafe or contraindicated
* Participants with central nervous system metastases will be excluded.
* Inability to comprehend and give informed consent

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mullinax, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Infusion of Tumor-infiltrating Lymphocyte: Participants will undergo tumor resection from which the tumor infiltrating lymphocyte (TIL) product will be generated. All participants will receive nonmyeloablative lymphodepleting chemotherapy with cyclophosphamide and fludarabine to enhance T-cell persistence and effectiveness in vivo. Cyclophosphamide will be administered at 60 mg/kg/day IV in 250 mL normal saline (NS). Fludarabine will then be infused at 25 mg/m^2 intravenous piggyback (IVPB). All participants will receive not less than 10^9, and up to 1x10^12 T cells in ≥250 mL NS as an inpatient by IV.
  Eight (8) to sixteen (16) hours after completing the T cell infusion, all participants will receive high-dose interleukin-2 (IL-2) on an inpatient basis at the standard dose of 600 000 IU/kg as an IV bolus over an approximate 15-minute period every 8 to 16 hours for up to 15 doses on days 1 to 5, as tolerated.
  TIL: Participants will receive an infusion of TIL after tumor resection and TIL product is generated.
  Interleukin-2 (IL-2): Participants will receive IL-2 600 000 IU/kg intravenously (IV) bolus (about 15 minutes) every 8 to 16 hours for up to 15 doses, beginning approximately 8 to 16 hours after T-cell infusion.
  Fludarabine: Participants will receive an IV infusion of Fludarabine 25 mg/m2 for approximately 30 minutes for 5 days, prior to T-Cell infusion
  Cyclophosphamide: Participants will receive Cyclophosphamide 60 mg/kg/day IV in 250 mL NS over approximately 2 hours, 7 days prior to T-Cell infusion
Period: Overall Study
Arm/Group | Infusion of Tumor-infiltrating Lymphocyte
Started | 9
Completed | 5
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Infusion of Tumor-infiltrating Lymphocyte
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Serious Adverse Events and Adverse Events
Description: Participants able to safely tolerate preparatory lymphodepletion, infusion of tumor-infiltrating lymphocytes (TIL) and subsequent IL-2, as measured by adverse events and serious adverse events.
Time Frame: Baseline to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion of Tumor-infiltrating Lymphocyte
Number analyzed (Participants) | 9
Participants
  Adverse event | 4
  No adverse events noted | 5

2. Secondary Outcome: Number of Participants With Objective Antitumor Response
Description: Number of participants with objective response (Complete Response (CR) + Progressive Response (PR)) rate at 12 weeks following TIL infusion, as measured by RECIST v1.1
Time Frame: At 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion of Tumor-infiltrating Lymphocyte
Number analyzed (Participants) | 9
Participants | 0

3. Secondary Outcome: Number of Participants With Circulating Tumor-infiltrating Lymphocytes (TIL) Product at 6 Weeks
Description: Number of participants with persistence of TIL infusion product at 6 weeks following treatment, as measured by T-cell receptor repertoire comparison between the infusion product and circulating Peripheral blood mononuclear cell (PBMC).
Time Frame: At 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion of Tumor-infiltrating Lymphocyte
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: 1 year
Description: AE's assessed at follow up visits.
Arm/Group | Infusion of Tumor-infiltrating Lymphocyte
All-Cause Mortality (participants affected / at risk) | 4/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infusion of Tumor-infiltrating Lymphocyte (N=9)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
General disorders and administration site conditions - Other, specify - Residual COVID-19 (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infusion of Tumor-infiltrating Lymphocyte (N=9)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (2)
Skin infection (Infections and infestations) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypotension (Vascular disorders) | 2 (3)
Encephalopathy (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT04052334/Prot_SAP_000.pdf